CLINICAL TRIAL: NCT05165498
Title: Reliability of Real-time Ultrasound Guidance as an Adjunct to Loss of Resistance for Thoracic Epidural Blocks
Brief Title: Real-time Ultrasound Guidance for Thoracic Epidural Blocks
Status: Not yet recruiting | Type: Observational
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Julian Aliste, Assistant Professor, University of Chile
Other Study IDs: OAIC 1037/19
Record Dates: First submitted 2021-12-07; First posted 2021-12-21 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Analgesia; Thoracic Tumors; Abdomen Tumors; Rib Fractures
Keywords: Thoracic peridural; Ultrasound-guided
MeSH Terms: conditions — Agnosia; Abdominal Neoplasms; Rib Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing elective thoracic surgery, abdominal surgery, or having rib fractures: Patients undergoing elective thoracic surgery, abdominal surgery, or having rib fractures who will have placed a thoracic epidural catheter to manage their perioperative analgesia.
  Interventions: Procedure: Real-time ultrasound guidance for thoracic epidural catheter placement.

INTERVENTIONS:
Procedure: Real-time ultrasound guidance for thoracic epidural catheter placement. — With an US-guided parasagittal oblique approach, the interlaminar space at the union between laminas and spinous processes at the predefined insertion level will be identified. A skin wheal will be raised with 3 mL of lidocaine 1%. Afterward, an 18-gauge Tuohy epidural block needle will be advanced under direct US vision until the tip is insinuated between the laminas and anchored to the flavum ligament. Then the needle will be attached to a low resistance syringe prefilled with saline solution and advanced until LOR to injection is confirmed. Then a 20-Gauge epidural catheter will be inserted 3-5 cm beyond the needle tip inside the epidural space and the needle removed.

SUMMARY:
Various modalities have been proposed for real-time confirmation of loss of resistance (LOR) for thoracic epidural blocks. With real-time ultrasound (US) guidance, the anesthesiologist attempts to visualize the sonographic advancement of the epidural needle and penetration of the epidural space (as detected by LOR)

This observational study is set out to confirm the reliability of real-time ultrasound guidance as an adjunct to LOR for thoracic epidural blocks.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* American Society of Anesthesiologists classification 1-3
* Body mass index between 20 and 35 (kg/m2)

Exclusion Criteria:

* Adults who are unable to give their own consent
* Sepsis (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. leukocytosis, increased c-reactive protein, increased procalcitonin)
* Coagulopathy (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. platelets ≤ 100, International Normalized Ratio ≥ 1.4 or prothrombin time ≥ 50)
* Allergy to local anesthetics (LAs)
* Prior surgery in the thoracic spine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective thoracic surgery, abdominal surgery, or suffering from rib fractures who will have placed a thoracic epidural catheter to manage their perioperative analgesia.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of successful epidural blocks after US-guided insertion of epidural catheters | 15 minutes after the local anesthetic injection through the epidural catheter
  After fifteen minutes of local anesthetic administration (4- mL dose of lidocaine 2% with epinephrine 5 μg/mL ), an investigator will apply ice to the T1 to L4 dermatomes bilaterally. The criterion standard for success will be the presence of an epidural block, defined as a block to ice in at least 2 dermatomes bilaterally. If operators could not advance the catheter past the needle tip after 2 attempts despite a 180-degree rotation of the bevel between the first and second attempts, epidural blocks will be considered failures.

SECONDARY OUTCOMES:
Number of blocked dermatomes | 15 minutes after the local anesthetic injection through the epidural catheter
  Number of blocked dermatomes after injection of local anesthetics through the epidural catheter.
Localization of blocked dermatomes | 15 minutes after the local anesthetic injection through the epidural catheter
  Localization of blocked dermatomes after injection of local anesthetics through the epidural catheter.
Image time | Up to 30 minutes after skin disinfection
  Needed time (minutes and seconds) to obtain an adequate image of the interlaminar space
Needle time | Up to 30 minutes after skin disinfection
  Needed time (minutes and seconds) to insert the Tuohy needle tip in the interlaminar space and confirm a loss of resistance
Catheter installation time | Up to 30 minutes after skin disinfection
  Elapsed time (minutes and seconds) from loss of resistance acquisition until the catheter is secured
Block performance time | Up to 30 minutes after skin disinfection
  Time (minutes and seconds) between skin disinfection and once the catheter is secured in place.
Epidural block-related complications | Up to 30 minutes after skin disinfection
  Incidence of adverse events related to epidural block or local anesthetic injection (i.e. paresthesia, accidental dural puncture, intravascular or subarachnoid position of catheters, intravascular, subarachnoid or subdural injection, local anesthetic systemic toxicity)

CONTACTS AND LOCATIONS:
Overall Officials: Julián Aliste, MD, Principal Investigator — University of Chile
Locations (1):
- Hospital Clínico Universidad de Chile, Santiago, Metropolitan, Chile

REFERENCES:
- [Background] Tran DQ, Van Zundert TC, Aliste J, Engsusophon P, Finlayson RJ. Primary Failure of Thoracic Epidural Analgesia in Training Centers: The Invisible Elephant? Reg Anesth Pain Med. 2016 May-Jun;41(3):309-13. doi: 10.1097/AAP.0000000000000394. PMID 27035462
- [Background] Tran DQ, Gonzalez AP, Bernucci F, Finlayson RJ. Confirmation of loss-of-resistance for epidural analgesia. Reg Anesth Pain Med. 2015 Mar-Apr;40(2):166-73. doi: 10.1097/AAP.0000000000000217. No abstract available. PMID 25642911
- [Background] Leurcharusmee P, Arnuntasupakul V, Chora De La Garza D, Vijitpavan A, Ah-Kye S, Saelao A, Tiyaprasertkul W, Finlayson RJ, Tran DQ. Reliability of Waveform Analysis as an Adjunct to Loss of Resistance for Thoracic Epidural Blocks. Reg Anesth Pain Med. 2015 Nov-Dec;40(6):694-7. doi: 10.1097/AAP.0000000000000313. PMID 26469364
- [Background] Arnuntasupakul V, Van Zundert TC, Vijitpavan A, Aliste J, Engsusophon P, Leurcharusmee P, Ah-Kye S, Finlayson RJ, Tran DQ. A Randomized Comparison Between Conventional and Waveform-Confirmed Loss of Resistance for Thoracic Epidural Blocks. Reg Anesth Pain Med. 2016 May-Jun;41(3):368-73. doi: 10.1097/AAP.0000000000000369. PMID 26894628
- [Background] Elgueta MF, Duong S, Finlayson RJ, Tran DQ. Ultrasonography for neuraxial blocks: a review of the evidence. Minerva Anestesiol. 2017 May;83(5):512-523. doi: 10.23736/S0375-9393.16.11650-5. Epub 2016 Nov 9. PMID 27827521
- [Background] Pak DJ, Gulati A. Real-Time Ultrasound-Assisted Thoracic Epidural Placement: A Feasibility Study of a Novel Technique. Reg Anesth Pain Med. 2018 Aug;43(6):613-615. doi: 10.1097/AAP.0000000000000761. PMID 29553999
- [Background] Yeager MP, Bae EE, Parra MC, Barr PA, Bonham AK, Sites BD. Fluoroscopy-assisted epidural catheter placement: an exploratory analysis of 303 pre-operative epidurograms. Acta Anaesthesiol Scand. 2016 Apr;60(4):513-9. doi: 10.1111/aas.12649. Epub 2015 Oct 28. PMID 26508378